CLINICAL TRIAL: NCT03173196
Title: Prospective Analysis of the Occurrence and Severity of Septic Encephalopathy in Patients With Severe Sepsis or Septic Shock, Including Non-invasive Multispectral Sonography
Brief Title: Prospective Analysis of Septic Associated Encephalopathy Using the Non-invasive Acoustocerebrography-ACG
Acronym: SAEACG
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Martin Sauer, MD, Deputy of the perioperative intensive care units, University of Rostock
Other Study IDs: A 2016-0026
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Encephalopathy; Organ Dysfunction Syndrome
Keywords: severe sepsis; encephalopathy
MeSH Terms: conditions — Brain Diseases; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sepsis group: Patients with a septic shock or a severe sepsis (surgical and non-surgical patients), staying on Intensive Care Unit, Non-invasive Multispectral Sonography - measurement
  Interventions: Device: Non-invasive Multispectral Sonography
- Non-septic group: Patients without sepsis (surgical and non-surgical patients), staying at least 24 hours on an Intensive Care Unit, Non-invasive Multispectral Sonography - measurement
  Interventions: Device: Non-invasive Multispectral Sonography

INTERVENTIONS:
Device: Non-invasive Multispectral Sonography — We measure both groups wirh the non-invasive multispectral sonography for 3 and for 30 minutes.

SUMMARY:
The patients of the group "sepsis" are measured several times with the non-invasive multi-spectral sonography (Sonovum "ACG-Diagnosesystem") (days 1, 3, 7 and 14). The patients of the group "control" are measured on days 1 and 3 with the system. A measurement takes 3 minutes. For this purpose two ultrasound heads are placed above the patient's ears and fixed with an all-head harness. The device is certified for CE application. There are no known health risks of ultrasound in humans.

DETAILED DESCRIPTION:
Sepsis with multiorgan failure is one of the most common diseases in intensive care units and is at the top of the world of causes of death. In addition to increasingly serious sepsis by multidrug-resistant pathogens, neurological symptoms are frequently recorded in the systemic manifestation of the disease pattern. Septic encephalopathy (SE) is usually an early cerebral sign of the developing sepsis, often before other clinically as well as diagnostically detectable findings such as fever ascent, hypotonia or laboratory chemical infections. Therefore, the SE is a clinically important parameter, also because after the sepsis, cerebral functional restrictions such as cognitive disorders can persist in the long term.

Therefore, on day 1, 3, 7 and 14 the patients are measured with the ACG-system as well as determined different scores of the patients: CAM-ICU (Confusion Assessment Method - Intensive Care Unit) and ICDSC (Intensive Care Delirium Screening Checklist) for the neurological outcome; Apache (Acute Physiology And Chronic Health Evaluation) II for mortality and SOFA (Sepsis-related Organ Failure Assessment Score) for organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock
* Clinical suspicion of septic encephalopathy
* consent to the study by the patient or legal representative
* stay in intensive care unit for at least 24 hours without the presence of a septic disease and without clinical guidance for an SE

Exclusion Criteria:

* Inability to consent to participation in the research project or rejection by patients or legal representatives
* existence of other causes of delir other than sepsis (e.g., withdrawal)
* Infrequent prognosis (expected death in ≤ 12 hours despite maximum therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * male or female, at least 18 years old
  * Severe sepsis or septic shock
  * Clinical suspicion of SE
  * consent to the study by the patient or legal representative
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Principal Components analysis vs ICDSC (Intensive Care Delirium Screening Checklist)-Score | Day 1
  after genetic algorithm to find two components
Principal Components analysis vs ICDSC / SOFA (Sepsis-related Organ Failure Assessment Score)-Score | Day 1
  after genetic algorithm to find two components

SECONDARY OUTCOMES:
ICDSC Score | Day 1
  Delirium Score: Intensive Care Delirium Screening Checklist
ICDSC Score | Day 3
  Delirium Score: Intensive Care Delirium Screening Checklist
SOFA Score | Day 1
  Organ Function Score: Sepsis-related Organ Failure Assessment Score
SOFA Score | Day 3
  Organ Function Score: Sepsis-related Organ Failure Assessment Score

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Units PIT 1+2, University Hospital Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sauer M, Sievert A, Wrobel M, Schmude P, Richter G. Acoustocerebrography in septic patients: A randomized and controlled pilot study. Front Med Technol. 2022 Sep 14;4:920674. doi: 10.3389/fmedt.2022.920674. eCollection 2022. PMID 36203789